CLINICAL TRIAL: NCT01532401
Title: Simplification of the Test of Sensibility in the Salt: Preliminary Study at the Child and the Adult
Brief Title: Oral Sodium Blood Pressure in Normal Weight, Overweight and Obese Volunteers
Acronym: PLADSEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PLADSEL 2010-023410-31
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2012-02

CONDITIONS: Obesity
Keywords: Blood pressure
MeSH Terms: conditions — Obesity | interventions — Sodium Chloride

ARMS (2):
- chlorure de sodium (Experimental)
  Interventions: Other: sodium chloride
- Methylcellulose (Placebo Comparator)
  Interventions: Other: Methylcellulose crystalline

INTERVENTIONS:
Other: sodium chloride — sodium chloride 500mg
  Arms: chlorure de sodium
Other: Methylcellulose crystalline — Methylcellulose 37 ml
  Arms: Methylcellulose

SUMMARY:
The primary objective of this study is to analyze the sensitivity of blood pressure to oral salt intake. Matched male and female participants will be selected as normal weight, overweight, and obese.

Participating subjects will have a first visit with blood pressure measurement and a blood sample. In two consecutive phases of one week, subjects will receive 12 pills of sodium (6 grams) or corresponding placebo. Blood pressure will be measured at the end of each phase.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18-45 for adults and 6-8 for children

Exclusion Criteria:

* African ethnicity (known to affect blood pressure sensitivity to salt)
* Chronic condition affecting blood pressure
* Diabetes (known to affect blood pressure sensitivity to salt)
* Hypertension

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samy HADJADJ, MD, Principal Investigator — CHU DE POITIERS-Service d'endocrinologie
Locations (1):
- Poitiers University Hospital, Poitiers, France